CLINICAL TRIAL: NCT01269333
Title: Impact of Omeprazole and Fluvoxamine on Platelet Response to Clopidogrel. a Randomized, Double-blind Placebo Controlled, Crossover Trial
Brief Title: Impact of Omeprazole and Fluvoxamine on Platelet Response to Clopidogrel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, RONNY ALCALAI, Cardiologist, Hadassah Medical Organization
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0330-HMO-CTIL
Record Dates: First submitted 2011-01-03; First posted 2011-01-04 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Drug Interaction of Clopidogrel
MeSH Terms: interventions — Omeprazole; Fluvoxamine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- fluvoxamine (Active Comparator)
  Interventions: Drug: fluvoxamine
- omeprazole (Experimental)
  Interventions: Drug: omeprazole
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: omeprazole — omeprazole 20mg for 7 days
  Arms: omeprazole
Drug: fluvoxamine — fluvoxamine 50mg for 7 days
  Arms: fluvoxamine
Drug: placebo — placebo for 7 days
  Arms: placebo

SUMMARY:
Clopidogrel is a platelets inhibitor that is widely used particularly during and after acute coronary events and coronary interventions. Several studies have shown that some patients are resistant to clopidogrel. The resistance mechanism is not entirely clear yet, but at least in part it is related to interactions between medications.

Omeprazole is a member in the family of gastric proton pump inhibitor (PPI) that are widely used in patients who receive combination of aspirin and clopidogrel in order to protect the stomach lining and prevent GI bleeding. Data from studies on platelet aggregation indicate that treatment with omeprazole may cause partial resistance to clopidogrel and increase risk for recurrent cardiovascular events in patients after coronary interventions. Recently the FDA published struck to avoid cross clopidogrel and omeprazole treatment for fear of reduction efficiency. Nevertheless there are several studies that do not support increased risk of cardiovascular events among patients taking omeprazole and clopidogrel, as the COGENT trial which is the single prospective controlled study that assessed the clinical implication of this drugs interaction.

The accepted Mechanism of interaction between omeprazole and clopidogrel is disturbance to create clopidogrel active metabolite through CYP2C19 inhibition by omeprazole. fluvoxamine - is a member in SSRIs family and a potent inhibitor of the CYP2C19. In vivo studies compared the degree of decomposition proguanil (a CYP2C19 indicator) by fluvoxamine and omeprazole found constant inhibition- Ki = 10 Micromol / L for of Omeprazole versus constant inhibition- Ki = 0.69 Micromol / L for fluvoxamine. This indicates a more potent inhibition of CYP2C19 in vivo of fluvoxamine compared to omeprazole. It is important to note that so far there is no date in literature studies demonstrates that there is any interaction between fluvoxamine and other CYP2C19 inhibitors and Clopidogrel.

Research goals:

* To assess the impact of fluvoxamine and omeprazole on platelet reactivity in healthy individuals treated with clopidogrel.
* To verify weather the mechanism of omeprazole-clopidogrel interaction is related to CYP2C19 inhibition.

Study design:

Randomized blinded placebo-controlled crossover trial on healthy volunteers. The response to clopidogrel will be assessed using two methods in subjects receiving clopidogrel and one of the study drugs: fluvoxamine, omeprazole or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Bleeding tendency

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2011-01; Primary Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
platlet reactivity in response to clopidogrel | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel